CLINICAL TRIAL: NCT03534661
Title: Role of a Nitric Oxide Synthase Inhibitor on GLP-2 Mediated Intestinal Lipoprotein Release
Brief Title: L-NMMA on GLP-2 Mediated Intestinal Lipoprotein Release
Acronym: LNMMA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: L-NMMA 13-6415
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2019-03

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — teduglutide; Saline Solution; omega-N-Methylarginine

STUDY DESIGN:
Intervention Model Description: Each participant receives 3 randomized treatments.
Who Masked: Participant
Masking Description: Single-blinded for participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teduglutide + Normal Saline (Placebo Comparator): Teguglutide + (L-NMMA control)
  Interventions: Drug: Teduglutide + Normal Saline
- Teduglutide + L-NMMA (Active Comparator): Tedulgutide + L-NMMA
  Interventions: Drug: Teduglutide + L-NMMA
- Placebo + L-NMMA (Placebo Comparator): (Teduglutide control) + L-NMMA
  Interventions: Drug: Placebo + L-NMMA

INTERVENTIONS:
Drug: Teduglutide + Normal Saline — Teduglutide 0.05 mg/kg subcutaneous injection; Normal Saline intravenous infusion
  Other Names: L-NMMA control
  Arms: Teduglutide + Normal Saline
Drug: Teduglutide + L-NMMA — Teduglutide 0.05 mg/kg subcutaneous injection; L-NMMA 10 mg/kg intravenous infusion
  Other Names: active treatments
  Arms: Teduglutide + L-NMMA
Drug: Placebo + L-NMMA — Placebo subcutaneous injection; L-NMMA 10 mg/kg intravenous infusion
  Other Names: Teduglutide control
  Arms: Placebo + L-NMMA

SUMMARY:
The gut is able to retain some fat for many hours after a fatty meal. The gut hormone glucagon-like peptide-2 (GLP-2) is known to release these fat stores in the gut, but it is not known how GLP-2 achieves this. One possibility is that GLP-2 increases blood flow in the gut. NG-monomethyl-L-arginine (L-NMMA) is a substance that inhibits nitric oxide synthase (an enzyme that helps make nitric oxide which increases blood flow). This protocol examines whether blocking gut blood flow with L-NMMA is able to prevent GLP-2 from releasing gut lipid stores. Healthy participants will be treated with a combination of Teduglutide (a resistant form of GLP-2) and L-NMMA, and their respective controls. Blood lipid levels will be measured following treatments.

DETAILED DESCRIPTION:
This is a single-blind, cross over, Phase 3b clinical study. The protocol aims to study 15 healthy, lean, non-diabetic males and females for three studies each, in random order, approximately four weeks apart, as follows.

Study A (L-NMMA + Teduglutide study): Volunteers will receive high-fat nutritional drink and seven hours later a subcutaneous injection of Teduglutide (0.05mg/kg of body weight, which is the FDA-approved route and daily dose for the treatment of short bowel syndrome).Thirty minutes prior to Teduglutide, the subject will receive an intravenous infusion of L-NMMA up to a maximum amount of 10 mg/kg, to inhibit nitric oxide synthesis. Lipid and lipoprotein levels will be measured at regular intervals for 3 hours following the injection of Teduglutide. Mesenteric blood flow will be measured at regular intervals by ultrasonography on some volunteers.

Study B (Teduglutide + normal saline): The design is identical to study A, except that, instead of L-NMMA, normal saline of the same volume will be infused.

Study C (Placebo + L-NMMA): The design is identical to study A, except that, instead of Teduglutide, a placebo will be injected subcutaneously.

Mesenteric Blood Flow measurement: Mesenteric blood flow will be measured at the bedside for some of the volunteers by ultrasonography in each study (A, B, C) before, during and after the administration of L-NMMA and Teduglutide. The first evaluation will begin 15 min before the start of the L-NMMA infusion and periodically afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 60 years
* Body mass index 20 kg/m2 to 30 kg/m2
* Hemoglobin above 130g/L.
* Normal glucose tolerance in response to a 75g, 2-hr oral glucose tolerance test

Exclusion Criteria:

* Subject has a history of hepatitis/hepatic disease that has been active within the previous two years.
* Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (creatinine > 1.5 mg/dL), genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic blood pressure > 100 or systolic > 180) or proliferative retinopathy
* History of diabetes or oral glucose tolerance indicative of diabetes or impaired glucose tolerance.
* Any history of a myocardial infarction or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on electrocardiogram, unstable angina, or decompensated heart failure.
* Any laboratory values: aspartate transaminase > 2x upper limit of normal; alanine aminotransferase > 2x upper limit of normal; thyroid-stimulating hormone > 6 miliunit/l
* Current addiction to alcohol or substances of abuse as determined by the investigator.
* Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
* Taking any prescription or non-prescription medications at the time of the study
* Having donated blood three months prior to and three months post study procedures
* A pregnancy test will be performed 1 to 3 days prior to each study in all female research participants. Those who test positive for pregnancy will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Plasma Lipid Levels | 10.5 hours
  Lipid levels in plasma and lipoprotein fractions are measured following treatments

SECONDARY OUTCOMES:
Blood Flow | 3 hours
  Mesenteric blood flow rates are measured with ultrasound following treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Tornto General Hospital, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No